CLINICAL TRIAL: NCT00129324
Title: Neurobehavioral Effects of Prevalent Neurotoxicants in Children: A Cohort Study of the Cincinnati Center for Children's Environmental Health
Brief Title: HOME Study (Health Outcomes and Measures of the Environment Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11261-CP-001; R01ES014575 (NIH); P01ES011261 (NIH); R01ES020349 (NIH); R01ES015517 (NIH); R01ES025214 (NIH); R01ES027224 (NIH); R01ES028277 (NIH); R01ES024381 (NIH); R01ES026903 (NIH); R01ES030078 (NIH); MDLTS0008-18 (Other Grant/Funding Number: HUD)
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Environmental Exposures; Child Development; Lead and Injury Reduction
Keywords: HOME; Environmental Exposure; Neurobehavior; Child Development; Lead Exposure; Child Injury; Adolescence; Adiposity; Neuroimaging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lead Reduction Arm (Other): random assignment to receive lead hazard control intervention. Assessing lead hazards in the home. Reducing lead hazards by cleaning, painting, covering, and/or replacing/repairing interior and exterior components of the home.
  Interventions: Procedure: Lead Hazard Control Intervention
- Injury Reduction Arm (Other): random assignment to receive injury hazard control intervention. Assessing home for potential injury hazards. Controlling hazards by 1) installing safety equipment such as stairway gates, cabinet locks, smoke & CO detectors, etc. 2) removing the hazards from the reach of a child and/or 3) restricting access to the hazards.
  Interventions: Procedure: Injury Hazard Control Intervention

INTERVENTIONS:
Procedure: Lead Hazard Control Intervention — Prior to their child's birth, participants randomized to Lead Reduction Group received lead hazard reduction controls to reduce residential exposure to lead.
  Arms: Lead Reduction Arm
Procedure: Injury Hazard Control Intervention — Between 3 and 6 months of age, participants randomized to Injury Reduction Arm received injury hazard controls to reduce the number of residential injuries.
  Arms: Injury Reduction Arm

SUMMARY:
The goal of the HOME Study is to quantify the impact of low-level fetal and early childhood exposures to environmental toxicants including lead, mercury, and other metals, pesticides, polychlorinated biphenyls (PCBs), persistent organic pollutants (PBDEs/PFCs), phthalates, phenols, environmental tobacco smoke, and alcohol on child development, neurobehavior, health, and growth. The HOME Study will also evaluate meconium as a biomarker for fetal exposure and test the effectiveness of home repairs to control lead hazards and injuries in early childhood.

DETAILED DESCRIPTION:
This study aims to examine the effects of low-level exposures to prevalent neurotoxicants on health, growth, and neurobehavior among a representative sample of children. Pregnant women were enrolled in the project around 16 weeks of gestation. In the first phase of the study, we followed children resulting from the pregnancy through the age of 36 months. The second phase extended follow-up through 72 months. Phase 3 extended follow-up to 8 years (range 7.5-10) with comprehensive neurobehavioral assessments. Phase 4 will allow follow-up at 12 years (range 11-13), and includes measures of health, growth and body composition, behavior and mental health, and neuroimaging. To address the potential adverse health risks of environmental chemicals, including persistent pollutants such as PBDEs and PFCs and other non-persistent chemicals, on fetal, infant, and child neurobehavior, the investigators are systematically examining their associations with endocrine function, cognition, learning and memory, motor skills, attention and executive function, and behavior from age 1 to 7.5-10 years. The investigators are also examining exposures at different developmental stages (in utero at 16 weeks of gestation, early childhood, school age, preadolescence) using stored biological samples and measure child neurobehavior at 1, 2, 3, 4, 5, 8, and 12 years. This longitudinal study will allow the investigators to determine the dose response, windows of susceptibility, and persistence of the association. The investigators are also examining the contribution of PBDE exposures from house dust in a subset of children who have complete sets of samples of maternal serum and child serum collected from annual visits along with extensive measures of mouthing behaviors.

Hypotheses from the four phases of the study are as follows:

1. In utero exposures measured by survey (alcohol and ETS), maternal and cord blood (lead and mercury) maternal and cord serum (ETS), and urine (pesticides) are less predictive of in utero effects of prevalent toxicants, including cognition, behavior problems, and growth compared with the same toxicants in meconium.
2. Prenatal and postnatal exposures to prevalent pesticides and ETS are associated with adverse neurobehavioral effects, and growth delay in children.
3. Higher lead exposure, measured during pregnancy and early childhood using maternal blood, cord blood, meconium and children's blood, will be associated with lower IQ scores and more behavioral problems for children with a maximal blood lead level < 5 mg/dL.
4. Children in the lead treatment arm will have: blood lead that is 2.7 mg/dL lower, higher IQ scores, greater growth velocity, and fewer behavioral problems than children in the control group.
5. Levels of lead in dust, soil and water will be significantly lower for housing units in the lead treatment arm compared with the injury control arm at 36 and 48 month home visits.
6. A multifactorial, housing intervention will reduce residential injury by 30 percent among children in the injury treatment arm compared with those in the lead treatment arm.
7. Prenatal and Postnatal exposures to PBDEs and PFCs are associated with altered thyroid hormone levels and deficits in infant and child neurobehavior
8. With increasing child age, PBDE exposure from household dust becomes a stronger predictor of child serum PBDE concentration than exposure from placenta or breast milk.
9. Developmental PBDE and PFC exposures are associated with internalizing symptoms.
10. Developmental PBDE and PFC exposures are associated with adverse changes in anatomical structure, neurochemistry, organization of white matter tracts, and connectivity of neural networks.
11. PFAS affect the gene expression and function of several biological pathways that program the fetus/infant towards a 'thrifty phenotype'. This leads to accelerated early childhood growth, increased fat mass, and features of metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Participating prenatal practice/clinic
* Participating hospital

Exclusion Criteria:

* Residence outside study area
* Plans to move outside study area within 1 year
* Home built after 1978
* Less than 18 years of age
* Beyond 19 weeks of gestation
* Diagnosis of diabetes
* Diagnosis of seizure disorder (taking anti-seizure medication)
* Diagnosis of thyroid disorder
* Diagnosis of AIDS or positive HIV test
* Diagnosis of bipolar disorder
* Diagnosis of schizophrenia
* Diagnosis of cancer resulting in radiation treatment or chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Lead reduction intervention, blood lead concentrations & neurobehavioral outcomes | 16wk & 26wk gestation, birth, annually at 1y-12y
  Testing the efficacy of lead reduction controls in the homes of participants. Examining the effects of low level blood lead concentration on child development and neurobehavior. Measures of blood lead concentration were taken from mothers prenatally at approximately 16 and 26 weeks gestation, from cord blood at birth, and annually from participating children from 1 - 10 years of age.
Exposure to environmental chemicals and their effects on child health, neurobehavior and development | 16wk & 26wk gestation, birth, 4wk postnatal, annually years 1-12.
  Addressing potential adverse health risks of environmental chemicals (persistent organic pollutants, metals, cotinine, pesticides, flame retardants, BPA, and phthalates) on fetal, infant, and child neurobehavior. Examining their associations with endocrine function, body composition (DXA), neuroimaging (MRI/fMRI), cognition, learning and memory, motor skills, attention and executive function, behavior, and mental health. Also examining exposures at different developmental stages and measuring child neurobehavior.
Injury prevention measures and household injuries | Postnatally up to age 5 years
  Test the efficacy of injury reduction controls in the homes of study participants. Assessed homes for potential injury hazards and installed child safety equipment. Collected parent report of injury events and validated the events against injuries tracked in the Hamilton County Injury Surveillance System

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Yolton, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Environmental Health Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Lanphear BP, Hornung R, Khoury J, Yolton K, Baghurst P, Bellinger DC, Canfield RL, Dietrich KN, Bornschein R, Greene T, Rothenberg SJ, Needleman HL, Schnaas L, Wasserman G, Graziano J, Roberts R. Low-level environmental lead exposure and children's intellectual function: an international pooled analysis. Environ Health Perspect. 2005 Jul;113(7):894-9. doi: 10.1289/ehp.7688. PMID 16002379
- [Background] Phelan KJ, Khoury J, Xu Y, Lanphear B. Validation of a HOME Injury Survey. Inj Prev. 2009 Oct;15(5):300-6. doi: 10.1136/ip.2008.020958. PMID 19805597
- [Background] Spanier AJ, Wilson S, Ho M, Hornung R, Lanphear BP. The contribution of housing renovation to children's blood lead levels: a cohort study. Environ Health. 2013 Aug 27;12:72. doi: 10.1186/1476-069X-12-72. PMID 23981571
- [Background] Braun JM, Kalloo G, Chen A, Dietrich KN, Liddy-Hicks S, Morgan S, Xu Y, Yolton K, Lanphear BP. Cohort Profile: The Health Outcomes and Measures of the Environment (HOME) study. Int J Epidemiol. 2017 Feb 1;46(1):24. doi: 10.1093/ije/dyw006. No abstract available. PMID 27006352
- [Background] Li N, Yolton K, Lanphear BP, Chen A, Kalkwarf HJ, Braun JM. Impact of Early-Life Weight Status on Cognitive Abilities in Children. Obesity (Silver Spring). 2018 Jun;26(6):1088-1095. doi: 10.1002/oby.22192. PMID 29797555
- [Background] Bowers K, Khoury J, Sucharew H, Xu Y, Chen A, Lanphear B, Yolton K. Early Infant Attention as a Predictor of Social and Communicative Behavior in Childhood. Int J Behav Dev. 2019 May;43(3):204-211. doi: 10.1177/0165025418797001. Epub 2018 Sep 18. PMID 37736344
- [Background] Goetz AR, Beebe DW, Peugh JL, Mara CA, Lanphear BP, Braun JM, Yolton K, Stark LJ. Longer sleep duration during infancy and toddlerhood predicts weight normalization among high birth weight infants. Sleep. 2019 Feb 1;42(2):zsy214. doi: 10.1093/sleep/zsy214. PMID 30412240
- [Background] Sears CG, Braun JM, Ryan PH, Xu Y, Werner EF, Lanphear BP, Wellenius GA. The association of traffic-related air and noise pollution with maternal blood pressure and hypertensive disorders of pregnancy in the HOME study cohort. Environ Int. 2018 Dec;121(Pt 1):574-581. doi: 10.1016/j.envint.2018.09.049. Epub 2018 Oct 6. PMID 30300815
- [Result] Geraghty SR, Khoury JC, Morrow AL, Lanphear BP. Reporting individual test results of environmental chemicals in breastmilk: potential for premature weaning. Breastfeed Med. 2008 Dec;3(4):207-13. doi: 10.1089/bfm.2008.0120. PMID 19086823
- [Result] Braun JM, Yolton K, Dietrich KN, Hornung R, Ye X, Calafat AM, Lanphear BP. Prenatal bisphenol A exposure and early childhood behavior. Environ Health Perspect. 2009 Dec;117(12):1945-52. doi: 10.1289/ehp.0900979. Epub 2009 Oct 6. PMID 20049216
- [Result] Braun JM, Daniels JL, Poole C, Olshan AF, Hornung R, Bernert JT, Khoury J, Needham LL, Barr DB, Lanphear BP. Prenatal environmental tobacco smoke exposure and early childhood body mass index. Paediatr Perinat Epidemiol. 2010 Nov;24(6):524-34. doi: 10.1111/j.1365-3016.2010.01146.x. Epub 2010 Aug 16. PMID 20955230
- [Result] Braun JM, Daniels JL, Poole C, Olshan AF, Hornung R, Bernert JT, Xia Y, Bearer C, Barr DB, Lanphear BP. A prospective cohort study of biomarkers of prenatal tobacco smoke exposure: the correlation between serum and meconium and their association with infant birth weight. Environ Health. 2010 Aug 27;9:53. doi: 10.1186/1476-069X-9-53. PMID 20799929
- [Result] Braun JM, Kalkbrenner AE, Calafat AM, Bernert JT, Ye X, Silva MJ, Barr DB, Sathyanarayana S, Lanphear BP. Variability and predictors of urinary bisphenol A concentrations during pregnancy. Environ Health Perspect. 2011 Jan;119(1):131-7. doi: 10.1289/ehp.1002366. PMID 21205581
- [Result] Wilson SE, Baker ER, Leonard AC, Eckman MH, Lanphear BP. Understanding preferences for disclosure of individual biomarker results among participants in a longitudinal birth cohort. J Med Ethics. 2010 Dec;36(12):736-40. doi: 10.1136/jme.2010.036517. Epub 2010 Oct 8. PMID 20935315
- [Result] Xu Y, Yolton K, Khoury J. Earliest appropriate time for administering neurobehavioral assessment in newborn infants. Pediatrics. 2011 Jan;127(1):e69-75. doi: 10.1542/peds.2010-1121. Epub 2010 Dec 20. PMID 21172999
- [Result] Braun JM, Kalkbrenner AE, Calafat AM, Yolton K, Ye X, Dietrich KN, Lanphear BP. Impact of early-life bisphenol A exposure on behavior and executive function in children. Pediatrics. 2011 Nov;128(5):873-82. doi: 10.1542/peds.2011-1335. Epub 2011 Oct 24. PMID 22025598
- [Result] Phelan KJ, Khoury J, Xu Y, Liddy S, Hornung R, Lanphear BP. A randomized controlled trial of home injury hazard reduction: the HOME injury study. Arch Pediatr Adolesc Med. 2011 Apr;165(4):339-45. doi: 10.1001/archpediatrics.2011.29. PMID 21464382
- [Result] Sathyanarayana S, Braun JM, Yolton K, Liddy S, Lanphear BP. Case report: high prenatal bisphenol a exposure and infant neonatal neurobehavior. Environ Health Perspect. 2011 Aug;119(8):1170-5. doi: 10.1289/ehp.1003064. Epub 2011 Apr 27. PMID 21524981
- [Result] Spanier AJ, Kahn RS, Xu Y, Hornung R, Lanphear BP. Comparison of biomarkers and parent report of tobacco exposure to predict wheeze. J Pediatr. 2011 Nov;159(5):776-82. doi: 10.1016/j.jpeds.2011.04.025. Epub 2011 Jun 8. PMID 21645908
- [Result] Spanier AJ, Kahn RS, Kunselman AR, Hornung R, Xu Y, Calafat AM, Lanphear BP. Prenatal exposure to bisphenol A and child wheeze from birth to 3 years of age. Environ Health Perspect. 2012 Jun;120(6):916-20. doi: 10.1289/ehp.1104175. Epub 2012 Feb 14. PMID 22334053
- [Result] Beebe DW, Rausch J, Byars KC, Lanphear B, Yolton K. Persistent snoring in preschool children: predictors and behavioral and developmental correlates. Pediatrics. 2012 Sep;130(3):382-9. doi: 10.1542/peds.2012-0045. Epub 2012 Aug 13. PMID 22891224
- [Result] Byars KC, Yolton K, Rausch J, Lanphear B, Beebe DW. Prevalence, patterns, and persistence of sleep problems in the first 3 years of life. Pediatrics. 2012 Feb;129(2):e276-84. doi: 10.1542/peds.2011-0372. Epub 2012 Jan 4. PMID 22218837
- [Result] Rauch SA, Braun JM, Barr DB, Calafat AM, Khoury J, Montesano AM, Yolton K, Lanphear BP. Associations of prenatal exposure to organophosphate pesticide metabolites with gestational age and birth weight. Environ Health Perspect. 2012 Jul;120(7):1055-60. doi: 10.1289/ehp.1104615. Epub 2012 Apr 5. PMID 22476135
- [Result] Sucharew H, Khoury JC, Xu Y, Succop P, Yolton K. NICU Network Neurobehavioral Scale profiles predict developmental outcomes in a low-risk sample. Paediatr Perinat Epidemiol. 2012 Jul;26(4):344-52. doi: 10.1111/j.1365-3016.2012.01288.x. Epub 2012 May 17. PMID 22686386
- [Result] Yolton K, Khoury J, Xu Y, Succop P, Lanphear B, Bernert JT, Lester B. Low-level prenatal exposure to nicotine and infant neurobehavior. Neurotoxicol Teratol. 2009 Nov-Dec;31(6):356-63. doi: 10.1016/j.ntt.2009.07.004. Epub 2009 Jul 17. PMID 19619640
- [Result] Yolton K, Xu Y, Strauss D, Altaye M, Calafat AM, Khoury J. Prenatal exposure to bisphenol A and phthalates and infant neurobehavior. Neurotoxicol Teratol. 2011 Sep-Oct;33(5):558-66. doi: 10.1016/j.ntt.2011.08.003. Epub 2011 Aug 10. PMID 21854843
- [Result] Braun JM, Kalkbrenner AE, Just AC, Yolton K, Calafat AM, Sjodin A, Hauser R, Webster GM, Chen A, Lanphear BP. Gestational exposure to endocrine-disrupting chemicals and reciprocal social, repetitive, and stereotypic behaviors in 4- and 5-year-old children: the HOME study. Environ Health Perspect. 2014 May;122(5):513-20. doi: 10.1289/ehp.1307261. Epub 2014 Mar 12. PMID 24622245
- [Result] Phelan KJ, Morrongiello BA, Khoury JC, Xu Y, Liddy S, Lanphear B. Maternal supervision of children during their first 3 years of life: the influence of maternal depression and child gender. J Pediatr Psychol. 2014 Apr;39(3):349-57. doi: 10.1093/jpepsy/jst090. Epub 2013 Dec 19. PMID 24357732
- [Result] Yolton K, Xu Y, Sucharew H, Succop P, Altaye M, Popelar A, Montesano MA, Calafat AM, Khoury JC. Impact of low-level gestational exposure to organophosphate pesticides on neurobehavior in early infancy: a prospective study. Environ Health. 2013 Sep 13;12(1):79. doi: 10.1186/1476-069X-12-79. PMID 24034442
- [Result] Braun JM, Lanphear BP, Calafat AM, Deria S, Khoury J, Howe CJ, Venners SA. Early-life bisphenol a exposure and child body mass index: a prospective cohort study. Environ Health Perspect. 2014 Nov;122(11):1239-45. doi: 10.1289/ehp.1408258. Epub 2014 Jul 29. PMID 25073184
- [Result] Braun JM, Froehlich T, Kalkbrenner A, Pfeiffer CM, Fazili Z, Yolton K, Lanphear BP. Brief report: are autistic-behaviors in children related to prenatal vitamin use and maternal whole blood folate concentrations? J Autism Dev Disord. 2014 Oct;44(10):2602-7. doi: 10.1007/s10803-014-2114-x. PMID 24710813
- [Result] Chen A, Yolton K, Rauch SA, Webster GM, Hornung R, Sjodin A, Dietrich KN, Lanphear BP. Prenatal polybrominated diphenyl ether exposures and neurodevelopment in U.S. children through 5 years of age: the HOME study. Environ Health Perspect. 2014 Aug;122(8):856-62. doi: 10.1289/ehp.1307562. Epub 2014 May 28. PMID 24870060
- [Result] Donauer S, Chen A, Xu Y, Calafat AM, Sjodin A, Yolton K. Prenatal exposure to polybrominated diphenyl ethers and polyfluoroalkyl chemicals and infant neurobehavior. J Pediatr. 2015 Mar;166(3):736-42. doi: 10.1016/j.jpeds.2014.11.021. Epub 2014 Dec 16. PMID 25524317
- [Result] Prasodjo A, Pfeiffer CM, Fazili Z, Xu Y, Liddy S, Yolton K, Savitz DA, Lanphear BP, Braun JM. Serum cotinine and whole blood folate concentrations in pregnancy. Ann Epidemiol. 2014 Jul;24(7):498-503.e1. doi: 10.1016/j.annepidem.2014.04.004. Epub 2014 Apr 24. PMID 24854185
- [Result] Spanier AJ, Kahn RS, Kunselman AR, Schaefer EW, Hornung R, Xu Y, Calafat AM, Lanphear BP. Bisphenol a exposure and the development of wheeze and lung function in children through age 5 years. JAMA Pediatr. 2014 Dec;168(12):1131-7. doi: 10.1001/jamapediatrics.2014.1397. PMID 25286153
- [Result] Watkins DJ, Eliot M, Sathyanarayana S, Calafat AM, Yolton K, Lanphear BP, Braun JM. Variability and predictors of urinary concentrations of phthalate metabolites during early childhood. Environ Sci Technol. 2014;48(15):8881-90. doi: 10.1021/es501744v. Epub 2014 Jul 9. PMID 24977926
- [Result] Kato K, Wong LY, Chen A, Dunbar C, Webster GM, Lanphear BP, Calafat AM. Changes in serum concentrations of maternal poly- and perfluoroalkyl substances over the course of pregnancy and predictors of exposure in a multiethnic cohort of Cincinnati, Ohio pregnant women during 2003-2006. Environ Sci Technol. 2014 Aug 19;48(16):9600-8. doi: 10.1021/es501811k. Epub 2014 Jul 29. PMID 25026485
- [Result] Barnard H, Rao R, Xu Y, Froehlich T, Epstein J, Lanphear BP, Yolton K. Association of the Conners' Kiddie Continuous Performance Test (K-CPT) Performance and Parent-Report Measures of Behavior and Executive Functioning. J Atten Disord. 2018 Sep;22(11):1056-1065. doi: 10.1177/1087054715578271. Epub 2015 Apr 6. PMID 25846228
- [Result] Braun JM, Chen A, Romano ME, Calafat AM, Webster GM, Yolton K, Lanphear BP. Prenatal perfluoroalkyl substance exposure and child adiposity at 8 years of age: The HOME study. Obesity (Silver Spring). 2016 Jan;24(1):231-7. doi: 10.1002/oby.21258. Epub 2015 Nov 11. PMID 26554535
- [Result] Romano ME, Webster GM, Vuong AM, Thomas Zoeller R, Chen A, Hoofnagle AN, Calafat AM, Karagas MR, Yolton K, Lanphear BP, Braun JM. Gestational urinary bisphenol A and maternal and newborn thyroid hormone concentrations: the HOME Study. Environ Res. 2015 Apr;138:453-60. doi: 10.1016/j.envres.2015.03.003. Epub 2015 Mar 17. PMID 25794847
- [Result] Vuong AM, Webster GM, Romano ME, Braun JM, Zoeller RT, Hoofnagle AN, Sjodin A, Yolton K, Lanphear BP, Chen A. Maternal Polybrominated Diphenyl Ether (PBDE) Exposure and Thyroid Hormones in Maternal and Cord Sera: The HOME Study, Cincinnati, USA. Environ Health Perspect. 2015 Oct;123(10):1079-85. doi: 10.1289/ehp.1408996. Epub 2015 Apr 17. PMID 25893858
- [Result] Werner EF, Braun JM, Yolton K, Khoury JC, Lanphear BP. The association between maternal urinary phthalate concentrations and blood pressure in pregnancy: The HOME Study. Environ Health. 2015 Sep 17;14:75. doi: 10.1186/s12940-015-0062-3. PMID 26380974
- [Result] Buckley JP, Engel SM, Braun JM, Whyatt RM, Daniels JL, Mendez MA, Richardson DB, Xu Y, Calafat AM, Wolff MS, Lanphear BP, Herring AH, Rundle AG. Prenatal Phthalate Exposures and Body Mass Index Among 4- to 7-Year-old Children: A Pooled Analysis. Epidemiology. 2016 May;27(3):449-58. doi: 10.1097/EDE.0000000000000436. PMID 26745610
- [Result] Engel SM, Bradman A, Wolff MS, Rauh VA, Harley KG, Yang JH, Hoepner LA, Barr DB, Yolton K, Vedar MG, Xu Y, Hornung RW, Wetmur JG, Chen J, Holland NT, Perera FP, Whyatt RM, Lanphear BP, Eskenazi B. Prenatal Organophosphorus Pesticide Exposure and Child Neurodevelopment at 24 Months: An Analysis of Four Birth Cohorts. Environ Health Perspect. 2016 Jun;124(6):822-30. doi: 10.1289/ehp.1409474. Epub 2015 Sep 29. PMID 26418669
- [Result] Xu Y, Khoury JC, Sucharew H, Dietrich K, Yolton K. Low-level gestational exposure to mercury and maternal fish consumption: Associations with neurobehavior in early infancy. Neurotoxicol Teratol. 2016 Mar-Apr;54:61-7. doi: 10.1016/j.ntt.2016.02.002. Epub 2016 Feb 12. PMID 26876455
- [Result] Harley KG, Engel SM, Vedar MG, Eskenazi B, Whyatt RM, Lanphear BP, Bradman A, Rauh VA, Yolton K, Hornung RW, Wetmur JG, Chen J, Holland NT, Barr DB, Perera FP, Wolff MS. Prenatal Exposure to Organophosphorous Pesticides and Fetal Growth: Pooled Results from Four Longitudinal Birth Cohort Studies. Environ Health Perspect. 2016 Jul;124(7):1084-92. doi: 10.1289/ehp.1409362. Epub 2015 Dec 18. PMID 26685281
- [Result] Donauer S, Altaye M, Xu Y, Sucharew H, Succop P, Calafat AM, Khoury JC, Lanphear B, Yolton K. An Observational Study to Evaluate Associations Between Low-Level Gestational Exposure to Organophosphate Pesticides and Cognition During Early Childhood. Am J Epidemiol. 2016 Sep 1;184(5):410-8. doi: 10.1093/aje/kwv447. Epub 2016 Aug 18. PMID 27539379
- [Result] Ehrhardt J, Xu Y, Khoury J, Yolton K, Lanphear B, Phelan K. Cognitive and motor abilities of young children and risk of injuries in the home. Inj Prev. 2017 Feb;23(1):16-21. doi: 10.1136/injuryprev-2016-042031. Epub 2016 Jul 19. PMID 27435102
- [Result] Percy Z, Xu Y, Sucharew H, Khoury JC, Calafat AM, Braun JM, Lanphear BP, Chen A, Yolton K. Gestational exposure to phthalates and gender-related play behaviors in 8-year-old children: an observational study. Environ Health. 2016 Aug 16;15(1):87. doi: 10.1186/s12940-016-0171-7. PMID 27527835
- [Result] Romano ME, Xu Y, Calafat AM, Yolton K, Chen A, Webster GM, Eliot MN, Howard CR, Lanphear BP, Braun JM. Maternal serum perfluoroalkyl substances during pregnancy and duration of breastfeeding. Environ Res. 2016 Aug;149:239-246. doi: 10.1016/j.envres.2016.04.034. Epub 2016 May 11. PMID 27179585
- [Result] Shoaff JR, Romano ME, Yolton K, Lanphear BP, Calafat AM, Braun JM. Prenatal phthalate exposure and infant size at birth and gestational duration. Environ Res. 2016 Oct;150:52-58. doi: 10.1016/j.envres.2016.05.033. Epub 2016 May 26. PMID 27236572
- [Result] Vuong AM, Braun JM, Sjodin A, Webster GM, Yolton K, Lanphear BP, Chen A. Prenatal Polybrominated Diphenyl Ether Exposure and Body Mass Index in Children Up To 8 Years of Age. Environ Health Perspect. 2016 Dec;124(12):1891-1897. doi: 10.1289/EHP139. Epub 2016 Jun 10. PMID 27285825
- [Result] Zhang H, Yolton K, Webster GM, Sjodin A, Calafat AM, Dietrich KN, Xu Y, Xie C, Braun JM, Lanphear BP, Chen A. Prenatal PBDE and PCB Exposures and Reading, Cognition, and Externalizing Behavior in Children. Environ Health Perspect. 2017 Apr;125(4):746-752. doi: 10.1289/EHP478. Epub 2016 Jul 6. PMID 27385187
- [Result] Vuong AM, Braun JM, Yolton K, Xie C, Webster GM, Sjodin A, Dietrich KN, Lanphear BP, Chen A. Prenatal and postnatal polybrominated diphenyl ether exposure and visual spatial abilities in children. Environ Res. 2017 Feb;153:83-92. doi: 10.1016/j.envres.2016.11.020. Epub 2016 Dec 1. PMID 27915227
- [Result] Braun JM, Bellinger DC, Hauser R, Wright RO, Chen A, Calafat AM, Yolton K, Lanphear BP. Prenatal phthalate, triclosan, and bisphenol A exposures and child visual-spatial abilities. Neurotoxicology. 2017 Jan;58:75-83. doi: 10.1016/j.neuro.2016.11.009. Epub 2016 Nov 23. PMID 27888119
- [Result] Vuong AM, Yolton K, Webster GM, Sjodin A, Calafat AM, Braun JM, Dietrich KN, Lanphear BP, Chen A. Prenatal polybrominated diphenyl ether and perfluoroalkyl substance exposures and executive function in school-age children. Environ Res. 2016 May;147:556-64. doi: 10.1016/j.envres.2016.01.008. Epub 2016 Jan 28. PMID 26832761
- [Result] Rosen-Carole CB, Auinger P, Howard CR, Brownell EA, Lanphear BP. Low-Level Prenatal Toxin Exposures and Breastfeeding Duration: A Prospective Cohort Study. Matern Child Health J. 2017 Dec;21(12):2245-2255. doi: 10.1007/s10995-017-2346-4. PMID 28735496
- [Result] Dasu K, Nakayama SF, Yoshikane M, Mills MA, Wright JM, Ehrlich S. An ultra-sensitive method for the analysis of perfluorinated alkyl acids in drinking water using a column switching high-performance liquid chromatography tandem mass spectrometry. J Chromatogr A. 2017 Apr 21;1494:46-54. doi: 10.1016/j.chroma.2017.03.006. Epub 2017 Mar 6. PMID 28336137
- [Result] Woods MM, Lanphear BP, Braun JM, McCandless LC. Gestational exposure to endocrine disrupting chemicals in relation to infant birth weight: a Bayesian analysis of the HOME Study. Environ Health. 2017 Oct 27;16(1):115. doi: 10.1186/s12940-017-0332-3. PMID 29078782
- [Result] Romano ME, Kalloo G, Etzel T, Braun JM. Re: Seasonal Variation in Exposure to Endocrine-disrupting Chemicals. Epidemiology. 2017 Sep;28(5):e42-e43. doi: 10.1097/EDE.0000000000000696. No abstract available. PMID 28570386
- [Result] Shoaff J, Papandonatos GD, Calafat AM, Ye X, Chen A, Lanphear BP, Yolton K, Braun JM. Early-Life Phthalate Exposure and Adiposity at 8 Years of Age. Environ Health Perspect. 2017 Sep 11;125(9):097008. doi: 10.1289/EHP1022. PMID 28935615
- [Result] Pell T, Eliot M, Chen A, Lanphear BP, Yolton K, Sathyanarayana S, Braun JM. Parental Concern about Environmental Chemical Exposures and Children's Urinary Concentrations of Phthalates and Phenols. J Pediatr. 2017 Jul;186:138-144.e3. doi: 10.1016/j.jpeds.2017.03.064. Epub 2017 May 2. PMID 28476460
- [Result] Millenson ME, Braun JM, Calafat AM, Barr DB, Huang YT, Chen A, Lanphear BP, Yolton K. Urinary organophosphate insecticide metabolite concentrations during pregnancy and children's interpersonal, communication, repetitive, and stereotypic behaviors at 8 years of age: The home study. Environ Res. 2017 Aug;157:9-16. doi: 10.1016/j.envres.2017.05.008. Epub 2017 May 11. PMID 28501654
- [Result] Stacy SL, Eliot M, Etzel T, Papandonatos G, Calafat AM, Chen A, Hauser R, Lanphear BP, Sathyanarayana S, Ye X, Yolton K, Braun JM. Patterns, Variability, and Predictors of Urinary Triclosan Concentrations during Pregnancy and Childhood. Environ Sci Technol. 2017 Jun 6;51(11):6404-6413. doi: 10.1021/acs.est.7b00325. Epub 2017 May 25. PMID 28516781
- [Result] Vuong AM, Yolton K, Xie C, Webster GM, Sjodin A, Braun JM, Dietrich KN, Lanphear BP, Chen A. Childhood polybrominated diphenyl ether (PBDE) exposure and neurobehavior in children at 8 years. Environ Res. 2017 Oct;158:677-684. doi: 10.1016/j.envres.2017.07.028. Epub 2017 Jul 19. PMID 28734254
- [Result] Stacy SL, Papandonatos GD, Calafat AM, Chen A, Yolton K, Lanphear BP, Braun JM. Early life bisphenol A exposure and neurobehavior at 8years of age: Identifying windows of heightened vulnerability. Environ Int. 2017 Oct;107:258-265. doi: 10.1016/j.envint.2017.07.021. Epub 2017 Jul 29. PMID 28764921
- [Result] Braun JM, Yolton K, Stacy SL, Erar B, Papandonatos GD, Bellinger DC, Lanphear BP, Chen A. Prenatal environmental chemical exposures and longitudinal patterns of child neurobehavior. Neurotoxicology. 2017 Sep;62:192-199. doi: 10.1016/j.neuro.2017.07.027. Epub 2017 Jul 20. PMID 28736150
- [Result] Zhang H, Yolton K, Webster GM, Ye X, Calafat AM, Dietrich KN, Xu Y, Xie C, Braun JM, Lanphear BP, Chen A. Prenatal and childhood perfluoroalkyl substances exposures and children's reading skills at ages 5 and 8years. Environ Int. 2018 Feb;111:224-231. doi: 10.1016/j.envint.2017.11.031. Epub 2017 Dec 20. PMID 29241079
- [Result] Kalloo G, Calafat AM, Chen A, Yolton K, Lanphear BP, Braun JM. Early life Triclosan exposure and child adiposity at 8 Years of age: a prospective cohort study. Environ Health. 2018 Mar 5;17(1):24. doi: 10.1186/s12940-018-0366-1. PMID 29506550
- [Result] Braun JM, Kalkwarf HJ, Papandonatos GD, Chen A, Lanphear BP. Patterns of early life body mass index and childhood overweight and obesity status at eight years of age. BMC Pediatr. 2018 May 11;18(1):161. doi: 10.1186/s12887-018-1124-9. PMID 29751833
- [Result] Jackson-Browne MS, Papandonatos GD, Chen A, Calafat AM, Yolton K, Lanphear BP, Braun JM. Identifying Vulnerable Periods of Neurotoxicity to Triclosan Exposure in Children. Environ Health Perspect. 2018 May 2;126(5):057001. doi: 10.1289/EHP2777. PMID 29727133
- [Result] Kingsley SL, Eliot MN, Kelsey KT, Calafat AM, Ehrlich S, Lanphear BP, Chen A, Braun JM. Variability and predictors of serum perfluoroalkyl substance concentrations during pregnancy and early childhood. Environ Res. 2018 Aug;165:247-257. doi: 10.1016/j.envres.2018.04.033. Epub 2018 May 7. PMID 29734025
- [Result] Romano ME, Eliot MN, Zoeller RT, Hoofnagle AN, Calafat AM, Karagas MR, Yolton K, Chen A, Lanphear BP, Braun JM. Maternal urinary phthalate metabolites during pregnancy and thyroid hormone concentrations in maternal and cord sera: The HOME Study. Int J Hyg Environ Health. 2018 May;221(4):623-631. doi: 10.1016/j.ijheh.2018.03.010. Epub 2018 Mar 23. PMID 29606598
- [Result] Li N, Arbuckle TE, Muckle G, Lanphear BP, Boivin M, Chen A, Dodds L, Fraser WD, Ouellet E, Seguin JR, Velez MP, Yolton K, Braun JM. Associations of cord blood leptin and adiponectin with children's cognitive abilities. Psychoneuroendocrinology. 2019 Jan;99:257-264. doi: 10.1016/j.psyneuen.2018.10.021. Epub 2018 Oct 25. PMID 30390444
- [Result] Braun JM, Hornung R, Chen A, Dietrich KN, Jacobs DE, Jones R, Khoury JC, Liddy-Hicks S, Morgan S, Vanderbeek SB, Xu Y, Yolton K, Lanphear BP. Effect of Residential Lead-Hazard Interventions on Childhood Blood Lead Concentrations and Neurobehavioral Outcomes: A Randomized Clinical Trial. JAMA Pediatr. 2018 Oct 1;172(10):934-942. doi: 10.1001/jamapediatrics.2018.2382. PMID 30178064
- [Result] Buck CO, Eliot MN, Kelsey KT, Calafat AM, Chen A, Ehrlich S, Lanphear BP, Braun JM. Prenatal exposure to perfluoroalkyl substances and adipocytokines: the HOME Study. Pediatr Res. 2018 Dec;84(6):854-860. doi: 10.1038/s41390-018-0170-1. Epub 2018 Sep 13. PMID 30250302
- [Result] Kalloo G, Wellenius GA, McCandless L, Calafat AM, Sjodin A, Karagas M, Chen A, Yolton K, Lanphear BP, Braun JM. Profiles and Predictors of Environmental Chemical Mixture Exposure among Pregnant Women: The Health Outcomes and Measures of the Environment Study. Environ Sci Technol. 2018 Sep 4;52(17):10104-10113. doi: 10.1021/acs.est.8b02946. Epub 2018 Aug 21. PMID 30088764
- [Result] Liang H, Vuong AM, Xie C, Webster GM, Sjodin A, Yuan W, Miao M, Braun JM, Dietrich KN, Yolton K, Lanphear BP, Chen A. Childhood polybrominated diphenyl ether (PBDE) serum concentration and reading ability at ages 5 and 8 years: The HOME Study. Environ Int. 2019 Jan;122:330-339. doi: 10.1016/j.envint.2018.11.026. Epub 2018 Nov 28. PMID 30503319
- [Result] Vuong AM, Braun JM, Webster GM, Thomas Zoeller R, Hoofnagle AN, Sjodin A, Yolton K, Lanphear BP, Chen A. Polybrominated diphenyl ether (PBDE) exposures and thyroid hormones in children at age 3 years. Environ Int. 2018 Aug;117:339-347. doi: 10.1016/j.envint.2018.05.019. Epub 2018 May 19. PMID 29787984
- [Result] Vuong AM, Braun JM, Yolton K, Wang Z, Xie C, Webster GM, Ye X, Calafat AM, Dietrich KN, Lanphear BP, Chen A. Prenatal and childhood exposure to perfluoroalkyl substances (PFAS) and measures of attention, impulse control, and visual spatial abilities. Environ Int. 2018 Oct;119:413-420. doi: 10.1016/j.envint.2018.07.013. Epub 2018 Jul 20. PMID 30015313
- [Result] Patel NB, Xu Y, McCandless LC, Chen A, Yolton K, Braun J, Jones RL, Dietrich KN, Lanphear BP. Very low-level prenatal mercury exposure and behaviors in children: the HOME Study. Environ Health. 2019 Jan 9;18(1):4. doi: 10.1186/s12940-018-0443-5. PMID 30626382
- [Derived] Nussbaumer-Streit B, Mayr V, Dobrescu AI, Wagner G, Chapman A, Pfadenhauer LM, Lohner S, Lhachimi SK, Busert LK, Gartlehner G. Household interventions for secondary prevention of domestic lead exposure in children. Cochrane Database Syst Rev. 2020 Oct 6;10(10):CD006047. doi: 10.1002/14651858.CD006047.pub6. PMID 33022752
- [Derived] Braun JM, Buckley JP, Cecil KM, Chen A, Kalkwarf HJ, Lanphear BP, Xu Y, Woeste A, Yolton K. Adolescent follow-up in the Health Outcomes and Measures of the Environment (HOME) Study: cohort profile. BMJ Open. 2020 May 7;10(5):e034838. doi: 10.1136/bmjopen-2019-034838. PMID 32385062
- See also: Related Info — https://www.cincinnatichildrens.org/research/divisions/g/pediatrics/labs/yolton